CLINICAL TRIAL: NCT02728141
Title: Timing, Duration and Severity of Infant Iron Deficiency: Developmental Impacts - Sucrose Component
Brief Title: Healthy Infant Development Project - Sucrose Component
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple
Other Study IDs: 1R01HD052069 (NIH)
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Iron Deficiency
MeSH Terms: conditions — Iron Deficiencies | interventions — Water; Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Water (Placebo Comparator): Newborn infants with ID numbers ending in odd numbers offered 2ml distilled water by syringe once in the side of the infant's mouth 2 minutes before heel stick.
  Interventions: Other: Water
- Sucrose (Active Comparator): Newborn infants with ID numbers ending in even numbers offered 2 ml 25% sucrose in distilled water by syringe once in the side of the infant's mouth 2 minutes before heel stick.
  Interventions: Other: Sucrose

INTERVENTIONS:
Other: Water — 2 ml distilled water by syringe one time in the newborn's mouth 2 minutes before heel stick
  Arms: Water
Other: Sucrose — 2 ml 25% sucrose in distilled water by syringe one time in the newborn's mouth 2 minutes before heel stick
  Arms: Sucrose

SUMMARY:
Iron deficiency affects the opioid and dopamine systems in rodent models, with a higher pain threshold. The opioid system is involved in sucrose's ability to reduce pain and distress during neonatal procedures. Thus, prenatal iron deficiency might affect response to pain and sucrose analgesia. In order to compare response to pain and sucrose during heel stick in neonates with and without iron deficiency, healthy full-term Chinese infants were randomized to receive sucrose or water by syringe beforehand, in conjunction with heel stick for metabolic screening.

ELIGIBILITY:
Inclusion Criteria:

* Full term healthy neonates participating in the Healthy Infant Development RCT (NCT00613717) in the folic acid/early postnatal placebo group and pre- and early postnatal iron-supplemented infants.

Exclusion Criteria:

* birth weight < 2500 g gestational age ≤ 37 wk major perinatal complications major congenital anomaly multiple birth

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 424 (Actual)
Dates: Start 2009-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Infant behavior (emotion regulation) | up to 5 days old
  Infant behavior observed included activity level, negative emotionality, alertness and soothability.

CONTACTS AND LOCATIONS:
Overall Officials: Betsy Lozoff, MD, Principal Investigator — University of Michigan
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
On request after main findings are published.

REFERENCES:
- [Derived] Lumeng JC, Li X, He Y, Gearhardt A, Sturza J, Kaciroti NA, Li M, Asta K, Lozoff B. Greater analgesic effects of sucrose in the neonate predict greater weight gain to age 18 months. Appetite. 2020 Mar 1;146:104508. doi: 10.1016/j.appet.2019.104508. Epub 2019 Nov 4. PMID 31698014